CLINICAL TRIAL: NCT00406224
Title: Effect of Oxygen Breathing on Flicker Induced Blood Flow Changes in the Optic Nerve Head
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FliOxyGen
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Healthy
MeSH Terms: interventions — Respiration; Oxygen

INTERVENTIONS:
Drug: breathing 100% oxygen

SUMMARY:
Background It has recently been shown that diffuse luminance flicker increases retinal and optic nerve head blood flow. This indicates that a neuro-vascular coupling between neural activity and blood flow exists as described previously for the brain. Although a lot of mediators such as NO, pO2, pCO2, H+ and K+ have been proposed, the mechanism of this coupling is still a matter of controversy. However, it has been shown in an animal experiment, that an increase in blood flow, evoked by diffuse luminance flicker stimulation is paralleled by an decrease in pO2 in the tissue. Thus, in this study we set out to investigate the flicker light induced increase in blood flow under elevated blood pO2.

Study rationale The motive for the investigation of retinal blood flow regulation is to enhance our understanding of the coupling mechanism between increased neural activity and blood flow in the retina in order to gain new insight in the pathophysiology of several eye diseases associated with ocular vascular disorders Study objectives To test the hypothesis whether oxygen breathing influences flicker light induced changes in optic nerve head blood flow

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Study Completion 2003-12

PRIMARY OUTCOMES:
Retinal vessel diameters

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhofer, MD, Principal Investigator — Medical University of Vienna